CLINICAL TRIAL: NCT07349108
Title: Comparison of Manual Vacuum Aspiration and Dilatation and Curettage for Endometrial Sampling Adequacy in Women With Abnormal Uterine Bleeding
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheikh Zayed Medical College (Other Government)
Responsible Party: Principal Investigator, Kainat usman, Principal Investigator, Sheikh Zayed Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sheikh ZMC/H3
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Abnormal Uterine Bleeding
Keywords: Abnormal uterine bleeding; Endometrial biopsy; Endometrial sampling; Endometrial tissue adequacy; Manual vacuum aspiration; Dilatation and curettage
MeSH Terms: conditions — Metrorrhagia; Dilatation, Pathologic | interventions — Dilatation and Curettage

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Manual Vacuum Aspiration (Experimental): Performed under paracervical block using 1% xylocaine with adrenaline in an outpatient setting.
  Interventions: Procedure: Manual Vacuum Aspiration
- Group Dilatation and Curettage (Active Comparator): Performed under paracervical block using 1% xylocaine with adrenaline.
  Interventions: Procedure: Dilatation and Curettage

INTERVENTIONS:
Procedure: Manual Vacuum Aspiration — Endometrial tissue was obtained using a handheld manual vacuum aspirator with appropriately sized cannula (No. 3 to No. 12), generating negative pressure to aspirate tissue from the endometrial cavity for histopathological examination.
  Arms: Group Manual Vacuum Aspiration
Procedure: Dilatation and Curettage — The cervix was gradually dilated using cervical dilators, followed by curettage of the endometrial lining with a curette to obtain tissue for histopathological examination.
  Arms: Group Dilatation and Curettage

SUMMARY:
This randomized controlled trial was conducted in the Department of Obstetrics and Gynecology, Sheikh Zayed Hospital, Rahim Yar Khan, to compare two commonly used methods for obtaining endometrial tissue in women aged 30 to 60 years presenting with abnormal uterine bleeding. Endometrial sampling is required to identify the underlying cause of abnormal bleeding, including precancerous changes and endometrial cancer. Participants who met eligibility criteria and provided informed consent were allocated to undergo either manual vacuum aspiration or dilatation and curettage. The primary purpose was to determine whether there was a significant difference between the two procedures in obtaining an adequate endometrial sample for histopathological reporting, where adequacy was defined as tissue containing both endometrial glands and stroma in sufficient quantity for interpretation. Pain severity was additionally assessed 24 hours after the procedure using a visual analog scale. The study hypothesis was that a significant difference existed in endometrial sampling adequacy between manual vacuum aspiration and dilatation and curettage among women with abnormal uterine bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 30-60 years.
* Patients presenting with abnormal uterine bleeding (AUB) as per operational definition.
* Patients who provide informed consent to participate in the study.

Exclusion Criteria:

* Patients with known pregnancy, active pelvic infection, or untreated sexually transmitted infections as per medical records.
* Patients with known coagulopathy, bleeding disorders, or currently on anticoagulant therapy.
* Patients with a history of endometrial or cervical cancer, abnormal Pap smear, pelvic pathology, or current hormonal use for endometrial pathology.
* Patients who have undergone surgical intervention involving the uterus in the past three months.
* Patients with severe medical conditions that could interfere with the study outcomes or pose a risk during the procedure (e.g., severe cardiovascular disease, uncontrolled diabetes).
* Patients with a history of severe allergic reactions to local anesthesia or NSAIDs were used in the study.
* Patients with stenotic cervical ostium.
* Females with malignancy undergoing chemotherapy or radiotherapy (as per medical records).

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females
Enrollment: 126 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Adequacy of endometrial tissue sample | During the procedure and at the time of histopathological examination of the collected specimen
  Adequacy of the endometrial specimen was determined by a consultant histopathologist and defined as the presence of both endometrial glands and stroma in at least 50% of the specimen, with minimal contamination by blood, mucus, or necrotic tissue, and preservation of tissue integrity sufficient for accurate histopathological interpretation.

SECONDARY OUTCOMES:
Post-procedure pain score | 24 hours after the endometrial sampling procedure
  Pain intensity was assessed using the Visual Analog Scale, a 10-centimeter scale ranging from 0 representing no pain to 10 representing the worst pain imaginable. Each participant marked the perceived pain level, and the recorded value was used for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Afshan Jabeen, Principal Investigator — Sheikh Zayed Medical college/Hospital, Rahimyar Khan
Locations (1):
- Sheikh Zayed Medical college/hospital, Rahim Yar Khan, Punjab Province, Pakistan